CLINICAL TRIAL: NCT00144586
Title: An Open-label, Extension, Phase III Study to Evaluate the Long-term Safety and Efficacy of MRA in Patients With RA Who Participated in Study MRA220JP or MRA221JP
Brief Title: Long-term Treatment Study of MRA for Rheumatoid Arthritis (RA) From Study MRA220JP or MRA221JP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRA222JP
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: MRA(Tocilizumab)

INTERVENTIONS:
Drug: MRA(Tocilizumab) — 8mg/kg/4 weeks

SUMMARY:
This is an open-label, extension, Phase III study to evaluate the long-term safety and efficacy of MRA in patients with RA who participated in Study MRA220JP or MRA221JP.

ELIGIBILITY:
Inclusion criteria

* RA patients who participated in the previous studies
* Patients who completed the last observation in the previous studies
* Patients who were confirmed to have no problems with safety in the previous studies.

Exclusion criteria

* Patients with Class IV Steinbrocker functional disorder at evaluation within 4 weeks before treatment with the investigational product
* Patients who were not enrolled by 3 months after the last observation day of the previous study

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2005-03; Primary Completion 2008-08 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
20% improvement based on the American College of Rheumatology (ACR) criteria compared with the baseline value in the previous study. | throughout study

SECONDARY OUTCOMES:
Time courses for DAS28, for ACR20%, 50%, and 70% improvement, and for each ACR core set variable. | Week 0, then every 4 Week

CONTACTS AND LOCATIONS:
Overall Officials: Yuji Kimura, Study Director — Chugai Pharmaceutical